CLINICAL TRIAL: NCT02364505
Title: Improving the Quality of Life of People With Multiple Sclerosis and Their Caregivers With a Telemedicine Mindfulness-Based Intervention
Brief Title: A Telemedicine Mindfulness-based Intervention for People With Multiple Sclerosis and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23042013205901
Record Dates: First submitted 2015-01-29; First posted 2015-02-18 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2016-01

CONDITIONS: Multiple Sclerosis
Keywords: caregivers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine mindfulness intervention (Experimental): Participants are assigned to a telemedicine mindfulness intervention group. The protocol lasts 8 weeks and it is composed by one online course session each week and home exercises. The course sessions, with a synchronous communication, will be conducted by a trainer, through teleconferences, that will explain how to practice the exercises to develop mindfulness attitude, following the mindfulness-based intervention-multiple sclerosis protocol. Subjects will be able to take part of these sessions everywhere, through a computer, tablet o mobile. During these sessions, individuals will interact with the trainer with teleconference or textual communications.
  Interventions: Behavioral: Telemedicine mindfulness-based intervention
- Psycho-education control group (Active Comparator): Psycho-education control group, provided with a telemedicine approach. Subject in this group will use a similar software than the experimental intervention, with identical time efforts required. Software contents will be psycho-educative.
  Interventions: Behavioral: Psycho-education intervention

INTERVENTIONS:
Behavioral: Telemedicine mindfulness-based intervention — Comparison of telemedicine mindfulness intervention with telemedicine psycho-education control group
  Arms: Telemedicine mindfulness intervention
Behavioral: Psycho-education intervention — Psycho-education control group, provided with a telemedicine approach. Subject in this group will use a similar software than the experimental intervention, with identical time efforts required. Software contents will be psycho-educative.
  Arms: Psycho-education control group

SUMMARY:
The aim of the project is to investigate the impact of a multiple sclerosis specific telemedicine mindfulness-based Intervention on the quality of life of people with multiple sclerosis and their caregivers.

DETAILED DESCRIPTION:
The mindfulness protocol will be modified according to multiple sclerosis clinical peculiarities and implemented with a multimedia web-based software.

The project will be divided in two parts. During the first phase of the project, a standard mindfulness-based stress reduction protocol will be modified according to clinical peculiarities and specific needs of people with multiple sclerosis. In the meanwhile, a multimedia software with these teaching will be developed, so that the training could be available online, from home. The protocol and the software will be tested for ergonomics in a pilot, qualitative, study.

In the second phase, a randomized clinical trial will be performed. One-hundred and twenty multiple sclerosis patients-caregivers couples will be randomly allocated in the experimental or to the control group. Subjects in the experimental group will attend the telemedicine mindfulness intervention, while controls will join a psycho-educational telemedicine program. At baseline, post-treatment and at a 6-month follow-up, participants will be assessed for quality of life, anxiety, depression, quality of sleep and mindfulness level. A subgroup of subjects will be assessed with actigraphs, for an objective evaluation of their sleep and physical activity. Experimental subjects will be assessed for participation and engagement to the treatment. Data will be analyzed with a complex longitudinal design, considering both within and between groups comparisons.

The dissemination process will involve scientific publication on neurological and psychological journals, a book, scientific meeting presentations and communication to general media. If there will be a positive effect of the mindfulness software, it will be diffused to multiple sclerosis clinics and associations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting or secondary progressive multiple sclerosis.
* Ability to communicate and to understand tasks.
* No change of disease-modifying treatment in the 3 months before the enrolment.
* No clinical relapses or use of steroid treatment during the 4 weeks before the enrolment.
* Availability of a personal computer, smartphone or tablet (compatible with the software).
* Provided informed consent for study participation.

Exclusion Criteria:

* Being a person who lives with the multiple sclerosis patient and provides him/her with most care and assistance
* Ability to communicate and to understand tasks
* Availability of a personal computer, smartphone or tablet (compatible with the software).
* Provided informed consent for study participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evidence of an improved quality of life in patients with multiple sclerosis as measured by The Multiple Sclerosis Quality of Life-54 (MSQOL-54) | First assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment
Evidence of an improved quality of life in caregivers as measured by the Short-Form-36 (SF-36) | First assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment
Evidence of a decrease of anxiety and depression in patients with multiple sclerosis and in caregivers as measured by the Hospital Anxiety and Depression Scale (HADS) | First assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment

SECONDARY OUTCOMES:
Evidence of an attained mindfulness level in patients with multiple sclerosis and in caregivers as measured by the Langer Mindfulness Scale (LMS) | first assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment
Evidence of a decrease of sleep disturbance and better quality of sleep in patients with multiple sclerosis and in caregivers as measured by the Medical Outcomes Study Sleep Measure (MOSssm) | First assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment
Evidence of a decrease of sleep disturbance and fatigue and a better quality of sleep in patients with multiple sclerosis as measured by actigraphy unit | First assessment includes the entires two weeks preceding the start of the intervention (baseline condition); second assessment includes the entire two weeks after the end of the intervention
  40 subjects will receive an actigraphy, a non-invasive method of monitoring human rest/activity cycles, that can be worn to measure gross motor activity
Evidence of a decrease in fatigue in patients with multiple sclerosis and in caregivers as measured by the Modified Fatigue Impact Scale (MFIS) | First assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment
Evidence of a decrease in caregiver burden as measured by the Zarit Burden Interview (ZBI) | First assessment: two weeks before the start of the intervention (baseline condition); second assessment: one week after the end of the intervention; third assessment: 6-months follow-up after the end of the intervention
  All subjects will be assigned to psychometric assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Pagnini, Milan, Mi, Italy

REFERENCES:
- [Background] Grossman P, Kappos L, Gensicke H, D'Souza M, Mohr DC, Penner IK, Steiner C. MS quality of life, depression, and fatigue improve after mindfulness training: a randomized trial. Neurology. 2010 Sep 28;75(13):1141-9. doi: 10.1212/WNL.0b013e3181f4d80d. PMID 20876468
- [Background] Whitebird RR, Kreitzer MJ, Lewis BA, Hanson LR, Crain AL, Enstad CJ, Mehta A. Recruiting and retaining family caregivers to a randomized controlled trial on mindfulness-based stress reduction. Contemp Clin Trials. 2011 Sep;32(5):654-61. doi: 10.1016/j.cct.2011.05.002. Epub 2011 May 12. PMID 21601010
- [Background] Teasdale JD, Segal Z, Williams JM. How does cognitive therapy prevent depressive relapse and why should attentional control (mindfulness) training help? Behav Res Ther. 1995 Jan;33(1):25-39. doi: 10.1016/0005-7967(94)e0011-7. PMID 7872934
- [Background] Manzoni GM, Pagnini F, Gorini A, Preziosa A, Castelnuovo G, Molinari E, Riva G. Can relaxation training reduce emotional eating in women with obesity? An exploratory study with 3 months of follow-up. J Am Diet Assoc. 2009 Aug;109(8):1427-32. doi: 10.1016/j.jada.2009.05.004. PMID 19631051
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Kraemer HC, Wilson GT, Fairburn CG, Agras WS. Mediators and moderators of treatment effects in randomized clinical trials. Arch Gen Psychiatry. 2002 Oct;59(10):877-83. doi: 10.1001/archpsyc.59.10.877. PMID 12365874
- [Background] Isaksson AK, Ahlstrom G. Managing chronic sorrow: experiences of patients with multiple sclerosis. J Neurosci Nurs. 2008 Jun;40(3):180-91. PMID 18578277
- [Background] Gay MC, Vrignaud P, Garitte C, Meunier C. Predictors of depression in multiple sclerosis patients. Acta Neurol Scand. 2010 Mar;121(3):161-70. doi: 10.1111/j.1600-0404.2009.01232.x. Epub 2010 Jan 12. PMID 20070277
- [Background] Feinstein A. Multiple sclerosis and depression. Mult Scler. 2011 Nov;17(11):1276-81. doi: 10.1177/1352458511417835. PMID 22058085
- [Background] Siegert RJ, Abernethy DA. Depression in multiple sclerosis: a review. J Neurol Neurosurg Psychiatry. 2005 Apr;76(4):469-75. doi: 10.1136/jnnp.2004.054635. PMID 15774430
- [Background] Riether AM. Anxiety in patients with multiple sclerosis. Semin Clin Neuropsychiatry. 1999 Apr;4(2):103-13. doi: 10.1053/SCNP00400103. PMID 10378954
- [Background] Mendozzi L, Tronci F, Garegnani M, Pugnetti L. Sleep disturbance and fatigue in mild relapsing remitting multiple sclerosis patients on chronic immunomodulant therapy: an actigraphic study. Mult Scler. 2010 Feb;16(2):238-47. doi: 10.1177/1352458509354551. Epub 2009 Dec 22. PMID 20028705
- [Background] Tachibana N, Howard RS, Hirsch NP, Miller DH, Moseley IF, Fish D. Sleep problems in multiple sclerosis. Eur Neurol. 1994;34(6):320-3. doi: 10.1159/000117070. PMID 7851452
- [Background] Sateia MJ, Nowell PD. Insomnia. Lancet. 2004 Nov 27-Dec 3;364(9449):1959-73. doi: 10.1016/S0140-6736(04)17480-1. PMID 15567013
- [Background] Buchanan RJ, Radin D, Chakravorty BJ, Tyry T. Informal care giving to more disabled people with multiple sclerosis. Disabil Rehabil. 2009;31(15):1244-56. doi: 10.1080/09638280802532779. PMID 19802928
- [Background] Pinquart M, Sorensen S. Differences between caregivers and noncaregivers in psychological health and physical health: a meta-analysis. Psychol Aging. 2003 Jun;18(2):250-67. doi: 10.1037/0882-7974.18.2.250. PMID 12825775
- [Background] Marziali E, Donahue P. Caring for others: Internet video-conferencing group intervention for family caregivers of older adults with neurodegenerative disease. Gerontologist. 2006 Jun;46(3):398-403. doi: 10.1093/geront/46.3.398. PMID 16731880
- [Background] Vitaliano PP, Zhang J, Scanlan JM. Is caregiving hazardous to one's physical health? A meta-analysis. Psychol Bull. 2003 Nov;129(6):946-72. doi: 10.1037/0033-2909.129.6.946. PMID 14599289
- [Background] Mitchell AJ, Benito-Leon J, Gonzalez JM, Rivera-Navarro J. Quality of life and its assessment in multiple sclerosis: integrating physical and psychological components of wellbeing. Lancet Neurol. 2005 Sep;4(9):556-66. doi: 10.1016/S1474-4422(05)70166-6. PMID 16109362
- [Background] Thomas PW, Thomas S, Hillier C, Galvin K, Baker R. Psychological interventions for multiple sclerosis. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004431. doi: 10.1002/14651858.CD004431.pub2. PMID 16437487
- [Background] Haase R, Schultheiss T, Kempcke R, Thomas K, Ziemssen T. Use and acceptance of electronic communication by patients with multiple sclerosis: a multicenter questionnaire study. J Med Internet Res. 2012 Oct 15;14(5):e135. doi: 10.2196/jmir.2133. PMID 23069209
- [Background] Boeschoten RE, Dekker J, Uitdehaag BM, Polman CH, Collette EH, Cuijpers P, Beekman AT, van Oppen P. Internet-based self-help treatment for depression in multiple sclerosis: study protocol of a randomized controlled trial. BMC Psychiatry. 2012 Sep 11;12:137. doi: 10.1186/1471-244X-12-137. PMID 22967202
- [Background] Akkus Y. Multiple sclerosis patient caregivers: the relationship between their psychological and social needs and burden levels. Disabil Rehabil. 2011;33(4):326-33. doi: 10.3109/09638288.2010.490866. Epub 2010 Jun 4. PMID 20521996
- [Background] Sorensen S, Pinquart M, Duberstein P. How effective are interventions with caregivers? An updated meta-analysis. Gerontologist. 2002 Jun;42(3):356-72. doi: 10.1093/geront/42.3.356. PMID 12040138
- [Background] Khalsa DS. Mindfulness effects on caregiver stress: should we expect more? J Altern Complement Med. 2010 Oct;16(10):1025-6. doi: 10.1089/acm.2010.0431. No abstract available. PMID 20954958
- [Background] Schulz R, Martire LM. Family caregiving of persons with dementia: prevalence, health effects, and support strategies. Am J Geriatr Psychiatry. 2004 May-Jun;12(3):240-9. PMID 15126224
- [Background] Winbush NY, Gross CR, Kreitzer MJ. The effects of mindfulness-based stress reduction on sleep disturbance: a systematic review. Explore (NY). 2007 Nov-Dec;3(6):585-91. doi: 10.1016/j.explore.2007.08.003. PMID 18005910
- [Background] Solari A, Filippini G, Mendozzi L, Ghezzi A, Cifani S, Barbieri E, Baldini S, Salmaggi A, Mantia LL, Farinotti M, Caputo D, Mosconi P. Validation of Italian multiple sclerosis quality of life 54 questionnaire. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):158-62. doi: 10.1136/jnnp.67.2.158. PMID 10406981
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Haigh EA, Moore MT, Kashdan TB, Fresco DM. Examination of the factor structure and concurrent validity of the Langer Mindfulness/Mindlessness Scale. Assessment. 2011 Mar;18(1):11-26. doi: 10.1177/1073191110386342. Epub 2010 Oct 27. PMID 20980699
- [Background] Hays RD, Martin SA, Sesti AM, Spritzer KL. Psychometric properties of the Medical Outcomes Study Sleep measure. Sleep Med. 2005 Jan;6(1):41-4. doi: 10.1016/j.sleep.2004.07.006. Epub 2004 Nov 11. PMID 15680294
- [Derived] Cavalera C, Rovaris M, Mendozzi L, Pugnetti L, Garegnani M, Castelnuovo G, Molinari E, Pagnini F. Online meditation training for people with multiple sclerosis: A randomized controlled trial. Mult Scler. 2019 Apr;25(4):610-617. doi: 10.1177/1352458518761187. Epub 2018 Feb 27. PMID 29485319
- [Derived] Cavalera C, Pagnini F, Rovaris M, Mendozzi L, Pugnetti L, Garegnani M, Molinari E. A telemedicine meditation intervention for people with multiple sclerosis and their caregivers: study protocol for a randomized controlled trial. Trials. 2016 Jan 4;17:4. doi: 10.1186/s13063-015-1136-9. PMID 26729330